CLINICAL TRIAL: NCT01297309
Title: A Long-term Open-label Study Investigating the Safety and Tolerability of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH[1-84]), for the Treatment of Adults With Hypoparathyroidism - A Clinical Extension Study (RACE)
Brief Title: A Open-label Study Investigating the Safety and Tolerability of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH [1-84]), for the Treatment of Adults With Hypoparathyroidism - A Clinical Extension Study (RACE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAR-C10-008
Record Dates: First submitted 2011-02-11; First posted 2011-02-16 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Hypoparathyroidism
Keywords: PTH 1-84; Hypoparathyroidism; Parathyroid Hormone 1-84; NPSP558
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPSP558 (Experimental): titration of 25, 50, 75 or 100 μg
  Interventions: Drug: NPSP558

INTERVENTIONS:
Drug: NPSP558 — All patients will inject NPSP558 individual titration of 25, 50, 75 or 100 μg SC QD into alternating thighs in the morning via a multidose injection pen device.
  Other Names: RACE

SUMMARY:
This study is a long-term, open-label study using NPSP558 for the treatment of adult patients with Hypoparathyroidism.

DETAILED DESCRIPTION:
Patients with a history of Hypoparathyroidism will be enrolled to receive study drug for up to 80 months, which will be injected daily in either thigh. During that time they will be monitored for safety (specifically calcium levels in blood or urine). In addition, the patients' intake of Vitamin D and Calcium will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Previously completed the rhPTH[1-84] RELAY study (8 weeks of active therapy) and/or previously completed the rhPTH[1-84] REPLACE study (Visit 18).
* Able to perform daily SC self-injections of study medication (or have a designee perform injection).
* Women who are (1) postmenopausal; (2) surgically sterilized; or, (3) of childbearing potential with a negative pregnancy test and who consent to use two acceptable methods of contraception for the duration of the study.
* Males who have female partners of childbearing potential must use two acceptable forms of contraception for the duration of the study.
* Serum creatinine <1.5 mg/dL at enrollment.
* Total serum calcium less than or equal to upper limit of normal (ULN) based on local laboratory result prior to enrollment.
* Serum 25 hydroxy (OH) vitamin D less than or equal to 1.5 times the ULN within approximately 16 weeks prior to enrollment.

Exclusion Criteria:

* Any condition that, in the investigator's opinion after consultation with the sponsor, would preclude the safe use of parathyroid hormone (PTH).
* Pregnant or lactating women.
* Any disease or condition which has a high probability of precluding the subject from completing the study or where the subject cannot or will not appropriately comply with study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-04-06 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (14):
  - Advance Medical Research LLC, Lakewood, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Bone & Mineral Clinic PC, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - University Physicians Group, Staten Island, New York
  - Physician East PA, Greenville, North Carolina
  - University of Cincinnati Bone Health and Osteoporosis Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cetero Research DGD Research Inc., San Antonio, Texas
  - The Vancouver Clinic, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ayodele O, Rejnmark L, Mu F, Lax A, Berman R, Swallow E, Gosmanova EO. Five-Year Estimated Glomerular Filtration Rate in Adults with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Nov;39(11):5013-5024. doi: 10.1007/s12325-022-02292-1. Epub 2022 Aug 26. PMID 36018496
- [Derived] Rejnmark L, Ayodele O, Lax A, Mu F, Swallow E, Gosmanova EO. The risk of chronic kidney disease development in adult patients with chronic hypoparathyroidism treated with rhPTH(1-84): A retrospective cohort study. Clin Endocrinol (Oxf). 2023 Apr;98(4):496-504. doi: 10.1111/cen.14813. Epub 2022 Aug 28. PMID 35974422
- [Derived] Ayodele O, Mu F, Berman R, Swallow E, Rejnmark L, Gosmanova EO, Kaul S. Lower Risk of Cardiovascular Events in Adult Patients with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Aug;39(8):3845-3856. doi: 10.1007/s12325-022-02198-y. Epub 2022 Jun 11. PMID 35696069
- [Derived] Chen KS, Gosmanova EO, Curhan GC, Ketteler M, Rubin M, Swallow E, Zhao J, Wang J, Sherry N, Krasner A, Bilezikian JP. Five-year Estimated Glomerular Filtration Rate in Patients With Hypoparathyroidism Treated With and Without rhPTH(1-84). J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3557-65. doi: 10.1210/clinem/dgaa490. PMID 32738041
- [Derived] Mannstadt M, Clarke BL, Bilezikian JP, Bone H, Denham D, Levine MA, Peacock M, Rothman J, Shoback DM, Warren ML, Watts NB, Lee HM, Sherry N, Vokes TJ. Safety and Efficacy of 5 Years of Treatment With Recombinant Human Parathyroid Hormone in Adults With Hypoparathyroidism. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5136-5147. doi: 10.1210/jc.2019-01010. PMID 31369089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 study centers in the United States between 06 April 2011 (first participant first visit) and 08 June 2018 (last participant last visit).
Pre-assignment Details: A total of 51 participants were enrolled and 49 participants received treatment out of them 37 participants completed the study.
Groups:
- rhPTH(1-84): Participants received rhPTH (1-84) subcutaneous injection with a starting dose of 25 or 50 microgram (mcg) once daily with dose adjusted by the investigator with upwards in increments of 25 mcg up to 100 mcg daily, with the goal to achieve or maintain total serum calcium levels in the range of 8.0 to 9.0 milligrams per deciliter (mg/dL).
Period: Overall Study
Arm/Group | rhPTH(1-84)
Started | 51
Treated | 49
Started Extension Period | 46
Completed | 37
Not Completed | 14
Not completed — Eligibility failure | 2
Not completed — Screen failure | 2
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 1
Not completed — Investigator Decision | 2
Not completed — Death | 1
Not completed — Participant not entering extensionperiod | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of study drug and had post baseline safety data.
Groups:
- rhPTH (1-84): Participants received rhPTH (1-84) subcutaneous injection with a starting dose of 25 or 50 microgram (mcg) once daily with dose adjusted by the investigator with upwards in increments of 25 mcg up to 100 mcg daily, with the goal to achieve or maintain total serum calcium levels in the range of 8.0 to 9.0 milligrams per deciliter (mg/dL).
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE) and Treatment Emergent Serious Adverse Event (TESAE)
Description: SAE is an adverse event (AE) that results in death, life threatening, persistent or significant incapacity or substantial disruption of ability to conduct normal life functions, hospitalization or prolongation of existing hospitalization, congenital anomaly or birth defect, important medical events that may not result in death, be life threatening, or require hospitalization. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical or medicinal product. Treatment emergent adverse events (TEAEs) were defined as AEs whose onset occurs, severity worsens or intensity increases after receiving the study medication of this study and <= 30 days after last dose of study drug.
Time Frame: From start of study drug administration up to follow-up (82 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Participants
  Number of participants with TESAE | 13
  Number of participants with TEAE | 48

2. Primary Outcome: Number of Responders With Calcium Source at Week 52
Description: A responder was defined as a participant who met all of the following 3 criteria at each (1) a greater than (>) 50% reduction from baseline or less than (<) 500 milligram (mg) of daily calcium supplementation. (2) a >50% reduction from baseline or <0.25 microgram (mcg) of daily calcitriol supplementation. (3) an albumin-corrected total serum calcium concentration that was normalized or maintained compared to the baseline greater than or equal to (>=) 1.875 millimoles per liter (mmol/L) and not exceeding the Upper Limit of Normal (ULN) values (2.15 to 2.55 mmol/L). End of Treatment (EOT) was defined as the last determination of response or last available measurement during the treatment period. Number of responders with calcium source for citrate and carbonate at week 52 was reported here.
Time Frame: Week 52
Population: ITT population included participants who received at least one dose of study drug and had at least one efficacy measurement. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 47
Participants
  Citrate (Responder): number analyzed (Participants) | 9
  Citrate (Responder) | 7
  Carbonate (Responder): number analyzed (Participants) | 28
  Carbonate (Responder) | 21

3. Primary Outcome: Number of Responders With Calcium Source at End Of Treatment (EOT) (Up to 82 Months)
Description: A responder was defined as a participant who met all of the following 3 criteria at each (1) a greater than (>) 50% reduction from baseline or less than (<) 500 milligram (mg) of daily calcium supplementation. (2) a >50% reduction from baseline or <0.25 microgram (mcg) of daily calcitriol supplementation. (3) an albumin-corrected total serum calcium concentration that was normalized or maintained compared to the baseline greater than or equal to (>=) 1.875 millimoles per liter (mmol/L) and not exceeding the Upper Limit of Normal (ULN) values (2.15 to 2.55 mmol/L). End of Treatment (EOT) was defined as the last determination of response or last available measurement during the treatment period. Number of responders with calcium source for citrate and carbonate at EOT was reported here.
Time Frame: EOT (up to 82 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 47
Participants
  Citrate (Responder): number analyzed (Participants) | 11
  Citrate (Responder) | 7
  Carbonate (Responder): number analyzed (Participants) | 29
  Carbonate (Responder) | 20

4. Secondary Outcome: Percent Change From Baseline in Oral Calcium Supplementation at Week 52 and EOT (Up to 82 Months)
Description: Percent change from baseline of oral calcium supplementation were reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, Week 52 and EOT (up to 82 months)
Population: ITT population included participants who received at least one dose of study drug and had at least one efficacy measurement.
Measure: Mean (Standard Deviation); unit: % change of oral calcium supplementation
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
% change of oral calcium supplementation
  Percent change from baseline at Week 52 | -68.7 (34.07)
  Percent change from baseline at EOT | -39.4 (107.23)

5. Secondary Outcome: Percent Change From Baseline in Oral Calcitriol Supplementation at Week 52 and EOT (Up to 82 Months)
Description: Percent change from baseline of oral calcitriol supplementation were reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, Week 52 and EOT (up to 82 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: %changeoforal calcitriol supplementation
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
%changeoforal calcitriol supplementation
  Percent change from baseline at Week 52 | -72.024 (44.6232)
  Percent change from baseline at EOT | -73.737 (39.3461)

6. Secondary Outcome: Percent Change From Baseline in Albumin Corrected Total Serum Calcium (ACSC) at EOT (Up to 82 Months)
Description: Percent change in ACSC was reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, EOT (up to 82 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change in ACSC
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Percent change in ACSC | -0.03 (0.190)

7. Secondary Outcome: Change From Baseline in 24-Hour Urine Calcium Excretion Through EOT (Up to 82 Months)
Description: Change in 24 hour urine calcium excretion was reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, EOT (up to 82 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimoles per day (mmol/day)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Millimoles per day (mmol/day)
  Baseline | 8.92 (5.009)
  Change from Baseline at EOT | -2.37 (5.809)

8. Secondary Outcome: Change From Baseline in 24-hour Urine Calcium Excretion in Participants Who Used Calcium-Sparing Diuretics Through EOT (Up to 82 Months)
Description: Change from baseline in urinary calcium concentration in participants who used at least one calcium-sparing diuretics and participants who not used calcium-sparing diuretics were reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, EOT (up to 82 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per day (mmol/day)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 47
Millimoles per day (mmol/day)
  EOT: Participants used calcium sparing diuretics: number analyzed (Participants) | 12
  EOT: Participants used calcium sparing diuretics | -4.07 (6.000)
  EOT:Participants without calcium sparing diuretics: number analyzed (Participants) | 35
  EOT:Participants without calcium sparing diuretics | -1.79 (5.713)

9. Secondary Outcome: Change From Baseline in Serum Calcium Concentration in Participants Who Used and Calcium Sparing Diuretics at EOT (Upto 82 Months)
Description: Change in serum calcium concentration of the number of participants who used at least one calcium-sparing diuretics and not used calcium sparing diuretics were reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, EOT (upto 82 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Millimoles per liter (mmol/L)
  EOT: Participants used calcium sparing diuretics: number analyzed (Participants) | 12
  EOT: Participants used calcium sparing diuretics | -0.21 (0.194)
  EOT:Participants without calcium sparing diuretics: number analyzed (Participants) | 37
  EOT:Participants without calcium sparing diuretics | -0.04 (0.200)

10. Secondary Outcome: Change From Baseline in Serum Phosphate at Month 72 and EOT (Upto 82 Months)
Description: Change of serum phosphate from baseline were reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, Month 72, EOT (upto 82 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per day (mmol/day)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Millimoles per day (mmol/day)
  Change from Baseline at Month 72: number analyzed (Participants) | 33
  Change from Baseline at Month 72 | -0.309 (0.2280)
  Change from Baseline at EOT | -0.254 (0.2924)

11. Secondary Outcome: Number of Participants Who Maintained a Calcium Phosphate Product in A Normal Range at EOT (Up to 82 Months)
Description: The normal range of calcium phosphate product is defined as <= 4.441 millimoles square per liter square (mmol^2/L^2).
Time Frame: EOT (up to 82 months)
Population: as for outcome 4
Measure: Number; unit: Count of participants
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Count of participants | 49

12. Secondary Outcome: Change From Baseline in Bone Turnover Markers at EOT (Up to 82 Months)
Description: Bone Turnover Markers such as bone specific alkaline phosphatase (BSAP), serum procollagen type 1 amino-terminal propeptide (P1NP) , osteocalcin were reported in particpiants. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, EOT (up to 82 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microgram per liter (μg/L)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
Microgram per liter (μg/L)
  EOT: Bone Specific alkaline phosphatase: number analyzed (Participants) | 47
  EOT: Bone Specific alkaline phosphatase | 5.27 (11.156)
  EOT: P1NP: number analyzed (Participants) | 48
  EOT: P1NP | 91.85 (104.327)
  EOT: Osteocalcin: number analyzed (Participants) | 47
  EOT: Osteocalcin | 10.06 (11.570)

13. Secondary Outcome: Change From Baseline in Serum Carboxy Terminal Telopeptide of Type I Collagen (s-CTx) Bone Turnover Marker at EOT (Up to 82 Months)
Description: Change form baseline in bone turnover marker (s-CTx)was reported. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, EOT (up to 82 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanogram per liter (ng/L)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 47
Nanogram per liter (ng/L) | 224.21 (295.858)

14. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) at Week 52 and EOT (Up to 82 Months)
Description: Change from baseline in BMD of lumbar spine (L1-L4), hip-total, hip-trochanter, hip-intertrochanter, hip-ward's triangle, hip-femoral neck, distal one third radius at Week 52 then every 12 months until EOT were assessed by dual-energy X-ray absorptiometry [DXA] and Z-score. EOT was defined as the last determination of response or last available measurement during the treatment period.
Time Frame: Baseline, Week 52 and EOT (up to 82 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram per square centimeter (g/cm^2)
Arm/Group | rhPTH (1-84)
Number analyzed (Participants) | 49
gram per square centimeter (g/cm^2)
  Lumbar Spine (L1-L4) - Change at Week 52: number analyzed (Participants) | 41
  Lumbar Spine (L1-L4) - Change at Week 52 | -0.0156 (0.0891)
  Lumbar spine (L1-L4) - Change at EOT: number analyzed (Participants) | 44
  Lumbar spine (L1-L4) - Change at EOT | -0.0272 (0.1111)
  Hip - Total - Change at Week 52: number analyzed (Participants) | 40
  Hip - Total - Change at Week 52 | -0.0189 (0.0572)
  Hip - Total - Change at EOT: number analyzed (Participants) | 43
  Hip - Total - Change at EOT | -0.0329 (0.0747)
  Hip - Femoral Neck - Change at Week 52: number analyzed (Participants) | 40
  Hip - Femoral Neck - Change at Week 52 | -0.0278 (0.0553)
  Hip - Femoral Neck - Change at EOT: number analyzed (Participants) | 43
  Hip - Femoral Neck - Change at EOT | -0.0364 (0.0848)
  Hip - Trochanter - Change at Week 52: number analyzed (Participants) | 40
  Hip - Trochanter - Change at Week 52 | -0.0235 (0.0542)
  Hip - Trochanter- Change at EOT: number analyzed (Participants) | 43
  Hip - Trochanter- Change at EOT | -0.0236 (0.1018)
  Hip - Ward's Triangle - Change at Week 52: number analyzed (Participants) | 40
  Hip - Ward's Triangle - Change at Week 52 | -0.0081 (0.0827)
  Hip - Ward's Triangle - Change at EOT: number analyzed (Participants) | 43
  Hip - Ward's Triangle - Change at EOT | -0.0178 (0.1014)
  Distal One Third Radius - Change at Week 52: number analyzed (Participants) | 41
  Distal One Third Radius - Change at Week 52 | -0.0006 (0.0629)
  Distal One Third Radius - Change at EOT: number analyzed (Participants) | 44
  Distal One Third Radius - Change at EOT | -0.0368 (0.0895)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Up to 82 months)
Description: Safety population included all participants who received at least one dose of study drug with any follow-up information and differ from the started population.
Arm/Group | rhPTH(1-84)
All-Cause Mortality (participants affected / at risk) | 2/49
Serious Adverse Events (participants affected / at risk) | 13/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhPTH(1-84) (N=49)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Biliary adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhPTH(1-84) (N=49)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (15)
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (42)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (17)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 (6)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Hot flush (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Colonic polyp (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 15 (20)
Paraesthesia oral (Gastrointestinal disorders) | 3 (5)
Toothache (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6)
Chest discomfort (General disorders) | 5 (5)
Fatigue (General disorders) | 8 (13)
Palpitations (Cardiac disorders) | 5 (5)
Seasonal allergy (Immune system disorders) | 3 (3)
Bronchitis (Infections and infestations) | 12 (16)
Cystitis (Infections and infestations) | 3 (3)
Ear infection (Infections and infestations) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 8 (12)
Herpes zoster (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 10 (11)
Nasopharyngitis (Infections and infestations) | 11 (22)
Sinusitis (Infections and infestations) | 16 (31)
Tooth infection (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (11)
Urinary tract infection (Infections and infestations) | 10 (14)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3)
Joint sprain (Injury, poisoning and procedural complications) | 7 (7)
Meniscus lesion (Injury, poisoning and procedural complications) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 6 (6)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Blood calcium decreased (Investigations) | 7 (7)
Blood glucose increased (Investigations) | 3 (3)
Urine calcium increased (Investigations) | 4 (9)
Vitamin D decreased (Investigations) | 5 (5)
Hypercalciuria (Renal and urinary disorders) | 5 (5)
Nephrolithiasis (Renal and urinary disorders) | 6 (9)
Renal cyst (Renal and urinary disorders) | 3 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 19 (50)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3)
Tetany (Metabolism and nutrition disorders) | 7 (40)
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 (8)
Dizziness (Nervous system disorders) | 7 (8)
Headache (Nervous system disorders) | 13 (22)
Hypoaesthesia (Nervous system disorders) | 3 (4)
Migraine (Nervous system disorders) | 4 (5)
Paraesthesia (Nervous system disorders) | 15 (32)
Tremor (Nervous system disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 7 (7)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (7):
  • Study Protocol: Original Protocol (2010-12-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/Prot_000.pdf
  • Study Protocol: Protocol Amendment 1 (2011-06-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/Prot_001.pdf
  • Study Protocol: Protocol Amendment 2 (2011-10-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/Prot_002.pdf
  • Study Protocol: Protocol Amendment 3 (2012-03-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/Prot_003.pdf
  • Study Protocol: Protocol Amendment 5 (2016-05-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/Prot_004.pdf
  • Study Protocol: Protocol Amendment 6 (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/Prot_005.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT01297309/SAP_006.pdf